CLINICAL TRIAL: NCT07380932
Title: Catheter Ablation for AF in Patients With Severe Mitral Regurgitation After Successful Transcatheter Mitral-Valve Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CABA-MiTRA-AFNET12
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Mitral Valve (MV) Regurgitation
Keywords: Atrial fibrillation; Mitral valve regurgitation; Mitral valve repair; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Gastroesophageal Reflux; Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: blinded endpoint assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other)
  Interventions: Other: Usual Care
- Pulmonary Vein Isolation (Other)
  Interventions: Other: Pulmonary Vein Isolation

INTERVENTIONS:
Other: Usual Care — Usual care will consist of optimal AF and heart failure therapy based on guideline recommendations and local protocols and usage. Individual treatment decisions will be taken by the site teams, considering the approved instruction for use (IFU) of medical devices and summary of product characteristics (SmPC) of all approved medications in patients with AF. The choice of therapies and medications follows routine care in line with medical guidelines and local policies at the discretion of the treating physician and should be based on the individual medical status of each study patient.
  Arms: Usual Care
Other: Pulmonary Vein Isolation — Patients randomised to AF ablation will undergo pulmonary vein isolation using a safe and effective technology within 30 days after randomisation.
  Arms: Pulmonary Vein Isolation

SUMMARY:
CABA-MiTRA-AFNET12 is a non-commercial, parallel-group, prospective, randomised, open, blinded endpoint assessment (PROBE), multi-centre, therapy strategy trial. The trial investigates patients with severe mitral valve regurgitation who have undergone transcatheter edge-to-edge mitral valve repair (M-TEER) and have concomitant atrial fibrillation (AF). The objective is to assess whether catheter ablation of AF is superior to standard-of-care treatment in patients after TEER in reduction of major adverse cardiovascular and cerebrovascular events (MACCE).

DETAILED DESCRIPTION:
The occurrence of atrial fibrillation (AF) as the most frequent arrhythmia is associated with an increased risk of stroke, acute coronary syndrome, heart failure, and cardiovascular death. AF is often associated with mitral valve regurgitation (MR) which represents the most frequent valvular heart disease in an elderly population. Both entities are not only linked by a complex pathophysiologic interplay but also the incidence of both is expected to increase due to the demographic factors, aging and obesity.

AF is also a frequent comorbidity in patients with mitral valve regurgitation (MR) undergoing transcatheter edge-to-edge repair (TEER) with an incidence between 33-53% in randomized controlled trials. This is of particular clinical relevance due the complex and deleterious interaction between AF, MR, and left ventricular dysfunction. AF may pronounce left ventricular systolic dysfunction and enhance functional MR by mitral annulus dilatation (3). Current data has shown that AF contributes markedly to the course of functional MR and determines an unfavourable outcome. Catheter ablation (CA) for AF in the setting of congestive heart failure (CHF) has recently been demonstrated to be associated with a prognostic benefit in all stages of systolic left ventricular heart failure (heart failure with reduced ejection fraction, HFrEF). Although, the benefit of rhythm control in general, but also after surgical mitral valve repair (MVR) has been shown data in the setting of AF in TEER is sparse. In a recent multi-center observational cohort, the outcome of patients undergoing CA before or after TEER was investigated. As a proof of concept, it was shown that CA was associated with a prognostic benefit outweighing the negative influence of AF. Thus, the present study aims at investigating the prognostic relevance of CA following TEER in a randomized, prospective design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented atrial fibrillation (AF).
* Transcatheter edge-to-edge mitral-valve repair (TEER) for severe functional mitral valve regurgitation (MR) with successful result (less than moderate MR, gradient < 5 mmHg) performed within a period of minimum of 30 days and a maximum of 6 months. Moderate residual MR is eligible if no further mitral valve intervention or surgery is planned and patient is stable for > 3 months.
* Provision of signed informed consent.

Exclusion Criteria:

* Age <18 years
* Patient not suitable for AF ablation
* Previous ablation procedure for AF
* Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular accident within 2 months prior to enrolment
* Untreated hypothyroidism or hyperthyroidism requiring therapy
* Enrolment in another randomised study
* Indication for cardiac resynchronization therapy
* Current pregnancy, breastfeeding, or women not using reliable contraceptive measures during fertility age
* Mental or physical inability to participate in the study
* Planned cardiovascular intervention or operation
* Life expectancy ≤ 12 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 956 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2031-07-01 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular complications related to AF | Throughout study completion, estimated at a median follow-up period of 33 months.
  It is defined as the time from randomisation to the first occurrence of (1) a composite of cardiovascular death, ischemic stroke or systemic embolic event,hospitalisation for heart failure (MACCE) and/or (2) death of any cause in a hierarchical order.
The Primary Safety Outcomes are the occurrence of AF ablation associated serious adverse events, hemorrhagic stroke, and non-serious adverse events of special interest. | Throughout study completion, estimated at a median follow-up period of 33 months.
  Serious Adverse Events (SAEs), including primary and secondary outcome parameters if based on clinical events, will be adjudicated by the independent Clinical Event Committee (CEC) according to standardised definitions given in the CEC charter.

SECONDARY OUTCOMES:
Time to individual components of first primary endpoint (MACCE) | Throughout study completion, estimated at a median follow-up period of 33 months.
Time to ECG or ILR documented AF recurrence | Throughout study completion, estimated at a median follow-up period of 33 months.
AF burden (ILR) assessed during the scheduled follow-up visits | Throughout study completion, estimated at a median follow-up period of 33 months.
Heart failure progression (pro-BNP) at 3 and 12 months compared to baseline | Throughout study completion, estimated at a median follow-up period of 33 months.
Heart failure progression (LV Function) at 3 and 12 months compared to baseline | Throughout study completion, estimated at a median follow-up period of 33 months
Heart failure progression (MR severity) at 3 and 12 months compared to baseline | Throughout study completion, estimated at a median follow-up period of 33 months
AF recurrence | Throughout study completion, estimated at a median follow-up period of 33 months.
Time to all-cause death | Throughout study completion, estimated at a median follow-up period of 33 months.
Time to cardiovascular death | Throughout study completion, estimated at a median follow-up period of 33 months.
Quality of life changes at 3 and 12 months compared to baseline (assessed by KCCQ-12) | Throughout study completion, estimated at a median follow-up period of 33 months.
Quality of life changes at 3 and 12 months compared to baseline (assessed by AFEQT) | Throughout study completion, estimated at a median follow-up period of 33 months.
Quality of life changes at 3 and 12 months compared to baseline (assessed by EQ-5D-5L) | Throughout study completion, estimated at a median follow-up period of 33 months.
  Quality of life as assessed by the EuroQol Group 5-Dimension 5-Level questionnaire (EQ-5D-5L): The resulting score of the UK index ranges from 1 (for the best state) to - 0.285 (for the worst state).
  EQ5D- VAS: visual-analogue scale (0 worst to 100 best).
Time to occurrence of atrial tachycardia(s) (ILR) | Throughout study completion, estimated at a median follow-up period of 33 months.
ECHO: LA size assessed as changes to baseline | Throughout study completion, estimated at a median follow-up period of 33 months.
ECHO: LA volume assessed as changes to baseline | Throughout study completion, estimated at a median follow-up period of 33 months.
ECHO: LV function assessed as changes to baseline | Throughout study completion, estimated at a median follow-up period of 33 months.
ECHO: MR grading assessed as changes to baseline | Throughout study completion, estimated at a median follow-up period of 33 months.
Time to AF progression (defined as change from paroxysmal to persistent AF as documented in the ILR) | Throughout study completion, estimated at a median follow-up period of 33 months.
Number of required of re-M-TEER procedures | Throughout study completion, estimated at a median follow-up period of 33 months.
Number of total ablations procedures | Throughout study completion, estimated at a median follow-up period of 33 months.
Number of nights spent in hospital (per year) | Throughout study completion, estimated at a median follow-up period of 33 months.
Any ablation other than the index procedure in the therapy arm. | Throughout study completion, estimated at a median follow-up period of 33 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Eckardt, MD, Study Director — University Hospital Münster; Daniel Steven, MD, Study Director — University Hospital Cologne; Reza Wakili, MD, Study Director — University Heart and Vascular Center Frankfurt; Stephan Willems, MD, Study Director — Asklepios Hospital St. Georg
Locations (4):
- Germany (4):
  - University Hospital Cologne, Cologne
  - University Heart and Vascular Center Frankfurt, Frankfurt
  - Asklepios Hospital St. Georg, Hamburg
  - University Hospital Münster, Münster